CLINICAL TRIAL: NCT06716866
Title: Temporally Interfering Electric Field Stimulation in the Treatment of Epilepsy - Effect of Temporal Interference on Biomarkers of Epilepsy
Brief Title: Temporally Interfering Electric Field Stimulation in the Treatment of Epilepsy
Acronym: EE-DES-TIEF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Emory University (Other); St. Anne's University Hospital Brno, Czech Republic (Other); Semmelweis University (Other); HÃ´pital de la Timone (MARSEILLE) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2042345
Record Dates: First submitted 2024-10-25; First posted 2024-12-04 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Epilepsy
Keywords: temporally-interfering electric fields
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Temporally-Interfering Electrical Field Central Nervous System Stimulation (Experimental): Participants in this arm receive temporally-interfering electric fields stimulation.
  Interventions: Device: temporally-interfering electric field stimulation

INTERVENTIONS:
Device: temporally-interfering electric field stimulation — Temporally-interfering electric field stimulation is a candidate non-invasive means to stimulate and modulate the nervous system. We do not know of any other trials of this method in epilepsy patients.
  Other Names: temporal interference electric field stimulation

SUMMARY:
This study investigates the potential for temporally-interfering electric field stimulation (TIEFS) to treat epilepsy. In this case series within and between subjects design, the impact of TIEFS on epilepsy biomarkers was studied in patients with medial temporal lobe epilepsy.

Secondary analyses examine the underlying physiological effects of TIEF on local brain activity and brain networks.

DETAILED DESCRIPTION:
Participants Patients with drug-resistant focal epilepsy and a clinical diagnosis of medial temporal epilepsy undergoing invasive intracranial electrophysiology studies will be consented in accord with institutional review boards at Emory University, Saint-Anne University Hospital, and the Institute of Neurosurgery and Neurointervention, Semmelweis University. The determination of medial temporal epilepsy is based on clinical semiology, EEG, PET, MRI, and invasive electrophysiology. Across all centers, patients underwent the stimulation protocols 6 to 10 days post-implantation after patient-specific electric field modeling to determine TIEFS electrode placement.

Patients then undergo two sessions of TIEFS on separate days, one sham (aligned carriers), and one active (with an offset in frequency between the carriers to provide a lower-frequency modulation envelope at the anatomical target.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing invasive intracranial EEG studies

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Reduction of Interictal Biomarkers of Epilepsy | From enrollment until the end of the admission for each patient (the admission is typically 7-14 days in duration).
  Three epilepsy interictal biomarkers will be examined: Interictal epileptiform discharges (IEDs), pathologic ripples (PRs), and high-frequency oscillations (HFOs). Each is recorded from intracranial field potential recordings (also 'intracranial electroencephalography' or iEEG). IEDs can also be recorded from scalp EEG where this is available (it is typically not recorded during iEEG studies). These features of the intracranial EEG will be measured at baseline, during sham TIEFS, and during active TIEFS.
  The primary outcome is the change in the number of IEDs during the baseline, sham, or active TIEFS periods. The secondary outcome is the number of PRs and HFOs during these periods.
  Semi-automated detection of IEDs, PRs, and HFOs will be performed using the freely available and validated AnyWave software ( INSERM and Aix-Marseille University) and its 'Delphos' detector. IEDs, PRs, and HFOs rates per minute will be determined.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - UC Davis Medical Center, Sacramento, California
  - Emory University Hospital, Atlanta, Georgia
- St. Anne Hospital, Masaryk University, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD will be shared with other researchers at the completion of the study.
  IPD in this study consists of the anatomical location of electrode contacts, electrophysiological recordings, field models of the carrier fields and interference envelope. IPD also includes neuroimaging, and key data from the clinical neurophysiology reports.
  All data will be fully de-identified.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: At the completion of the studies.
Access Criteria: Data will be shared upon request to the investigative team for non-commercial and academic use.